CLINICAL TRIAL: NCT07264387
Title: Predictive Factors for Return to Work After a First Stroke Treated at Clermont-Ferrand University Hospital in Puy de Dôme Between January 2020 and December 2024
Acronym: RTWS2
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2025 ORANGE
Record Dates: First submitted 2025-09-12; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Stroke
Keywords: stroke; return to work; predictive factors
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Stroke is a leading cause of acquired motor disability and the second most common cause of major cognitive impairment worldwide. In France, approximately 150,000 new cases occur annually, with around 31% affecting individuals of working age, making return to work (RTW) a critical public health issue. Beyond the medical burden, stroke has profound socio-economic consequences, including loss of productivity, prolonged sick leave, part-time resumption, and the need for workplace adaptations. While RTW after stroke has been investigated, major gaps remain. No standardized recommendations exist for vocational reintegration, and predictive factors are still debated. Quantitative determinants such as stroke type, severity, functional independence, and occupational characteristics have been identified, but qualitative aspects-including self-efficacy, perceived social burden, employer relationships, and motivation-are poorly documented. Moreover, cognitive deficits are often insufficiently characterized, as screening tools such as MMSE or MoCA lack the sensitivity of comprehensive neuropsychological assessments. The impact of revascularization procedures on RTW and the ability to sustain employment after initial resumption also remain unclear. Importantly, no recent data are available in the Auvergne region, despite evolving labor policies that may influence reintegration trajectories. This observational study therefore aims to identify both quantitative and qualitative predictors of RTW after ischemic or hemorrhagic stroke, describe vocational pathways in a regional cohort, and explore barriers and facilitators to long-term reintegration. Ultimately, the study seeks to provide updated evidence to guide tailored rehabilitation and socio-professional reintegration strategies, supporting sustainable RTW in working-age stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have suffered an ischaemic stroke according to ICD-10 (ICD-10 code: I63 (cerebral infarction) I64 (unspecified stroke), I69 (sequelae of cerebrovascular disease) or patients who have had a haemorrhagic stroke according to ICD-10 (ICD-10 code: I60, I61 and I62) between January 2020 and March 2024
* Patients of working age/under 64 years of age (legal retirement age)
* Patients with an employment contract at the time of the stroke
* Patients treated at Clermont-Ferrand University Hospital
* Post-stroke consultation recorded in the patient's medical file
* Patients affiliated with the social security system
* Patients who have not objected to participating in the study

Exclusion Criteria:

* Patients with a history of ischaemic or haemorrhagic stroke
* Patients with a history of head trauma with neurological sequelae corresponding to codes S060, S061, S062, S063, S065, S066, S067, S068 and S069
* Patients who died as a result of stroke
* Patients unable to respond to telephone questionnaires
* Patients under guardianship or trusteeship
* Patients who have suffered a transient ischaemic attack (TIA) (G459 according to ICD 10)
* Patients who were in early retirement at the time of assessment
* No information on employment after stroke in the medical file
* Patients with category 2 or 3 disability prior to stroke due to another condition
* Patients on sick leave prior to stroke due to another condition
* Patients receiving RSA income support

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Stroke management follows a continuum, starting with acute care in neurology and neurosurgery, then progressing to medium- and long-term multidisciplinary rehabilitation in the Physical Medicine and Rehabilitation (PMR) department of Clermont-Ferrand University Hospital. Within this context, return to work is a key objective, supported by the expertise of PMR teams and close collaboration with neurology and neurosurgery. To conduct this study, authorisation to access medical records was granted by the Medical Information Department (DIM), covering patients under 64 years old admitted for ischaemic or haemorrhagic stroke between January 2020 and December 2024. Screening will be performed on hospitalisations in neurology and neurosurgery, and all eligible patients experiencing a first stroke during this period will be invited to participate.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Return to work rate | At inclusion
  Percentage of return to work after a first ischaemic or haemorrhagic stroke between January 2020 and December 2024 in patients of working age.
Factors correlated with return to work | At inclusion
  Determine the factors associated with return to work (gender)
Factors correlated with return to work | At inclusion
  Determine the factors associated with return to work (stroke severity)
Factors correlated with return to work | At inclusion
  Determine the factors associated with return to work (stroke type (ischaemic or haemorrhagic)).
Factors correlated with return to work | At inclusion
  Determine the factors associated with return to work (independence)
Factors correlated with return to work | At inclusion
  Determine the factors associated with return to work (occupation)

SECONDARY OUTCOMES:
Quality of life after stroke | At inclusion
  The Short-Form-12 (SF-12) questionnaire is a standardized self-administered questionnaire used to assess health-related quality of life. It comprises 12 questions covering 8 domains: physical activities, physical and mental limitations, pain, perceived general health, vitality, mental health and social relationships. Each item is rated on a 5- or 6-point Likert scale. The responses are used to calculate two scores: a physical composite score (PCS) and a mental composite score (MCS), each ranging from 0 (perceived health status very poor) to 100 (perceived health status optimal).
Anxiety and Depression scale | At inclusion
  The Hospital Anxiety and Depression Scale (HADs) questionnaire is a psychometric self-assessment questionnaire consisting of 14 items divided into two subscales (anxiety and depression) of seven items each. Each item is rated on a scale of 0 to 3. A score is given for each subscale, A for anxiety and D for depression. The score can range from 0 (no anxiety and/or depressive disorders) to 21 (proven anxiety and/or depressive disorders of varying severity) for each subscale.
Fatigue Severity Scale | At inclusion
  The Fatigue Severity Scale (FSS) questionnaire is a self-assessment tool used to evaluate the severity of fatigue and its impact on daily activities. This questionnaire consists of nine items rated on a seven-point Likert scale, ranging from 1 ('strongly disagree') to 7 ('strongly agree'). The score ranges from 7 (no fatigue in daily activities) to 63 (extreme fatigue in daily activities). A score above 36 indicates that the patient may need to have their fatigue assessed by a healthcare professional.
Predictive score for return-to-work rate | At inclusion
  Develop a predictive score for return to work using the predictive factors for return to work identified in the main objective.
Job retention | At inclusion
  To study job retention and its association with factors such as stroke severity.

CONTACTS AND LOCATIONS:
Overall Officials: Lise Laclautre, Study Director — University Hospital, Clermont-Ferrand
Locations (2):
- France (2):
  - Clermont Ferrand University Hospital, Louise Michel site, Cébazat, France
  - CHU Clermont-Ferrand, Louise Michel, Clermont-Ferrand

IPD SHARING:
Plan to Share IPD: No